CLINICAL TRIAL: NCT01323907
Title: Compassionate Use of Omegaven IV Fat Emulsion in Infants With Life Threatening Parenteral Nutrition-associated Liver Disease (PNALD).
Brief Title: Compassionate Use of Omegaven IV Fat Emulsion
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Omegaven is now FDA approved.
Sponsor: Sivan Kinberg (Other)
Responsible Party: Sponsor-Investigator, Sivan Kinberg, Assistant Professor of Pediatrics at the Columbia University Medical Center, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAF2546
Record Dates: First submitted 2011-03-16; First posted 2011-03-28 (Estimated); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Total Parenteral Nutrition-induced Cholestasis
Keywords: Total Parenteral Nutrition-induced Cholestasis; Omegaven; liver disease; Cholestasis; Fat emulsions
MeSH Terms: conditions — Liver Diseases; Cholestasis | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Omegaven (Experimental): Omegaven IV lipid emulsion administration for infants with life threatening parenteral nutrition associated liver disease
  Interventions: Drug: Omegaven IV lipid emulsion

INTERVENTIONS:
Drug: Omegaven IV lipid emulsion — For infants meeting inclusion criteria and whose guardians consent to participation, Omegaven will be initiated at the dose of 0.5gram/kg/day and is infused over 24 hours for 1-2 days and then advanced to 1 gram/kg/day. Omegaven will be infused intravenously through a central or peripheral catheter alone or in conjunction with parenteral nutrition.
  Other Names: Omega-3 Fatty Acids

SUMMARY:
The purpose of the study is to provide use of Omegaven in children with life threatening Total Parenteral Nutrition (TPN) associated cholestasis when all other medical and surgical treatments/therapies have been either ineffective or not feasible in the treatment of this serious condition. This is a compassionate use protocol.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of life threatening PNALD
* Dependent on Parenteral Nutrition for caloric needs
* Expected to require PN for at least another 30 days
* Other causes of liver disease have been excluded
* GI/Liver service is involved in patient care
* Standard therapies for the treatment of PNALD must have been utilized prior to initiating omegaven.
* Inpatient at Morgan Stanley Children's Hospital of NewYork Presbyterian Hospital
* Must be at least 2 months of age

Exclusion Criteria:

* Not inpatient
* Younger than 2 months of age
* Expected to be weaned off of parenteral nutrition within 30 days
* have other documented causes of liver disease
* have signs of proven severe advanced liver disease
* Allergy to seafood, egg protein and/or previous allergy to Omegaven
* active coagulopathy, impaired lipid metabolism or severe hyperlipidemia with or without pancreatitis, stoke, embolism, hemodynamic collapse or shock, recent MI, cholestasis due to any reason other than PNALD, active new infection at time of initiation of Omegaven, hemodynamic instability or if unable to tolerate the necessary laboratory monitoring
* must not be enrolled in another clinical trial involving an investigational agent (unless approved by the designated physicians).
* Parent or legal guardian must be willing to provide consent.

Ages: 2 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2011-01 (Estimated); Primary Completion 2019-02-13 (Actual); Study Completion 2019-02-13 (Actual)

PRIMARY OUTCOMES:
Reduction of direct serum bilirubin level (mg/dL) | Up to 6 months from the completion of the study.
  For effectiveness endpoint, the allowable minimum time interval between serial direct bilirubin measurements that will determine reversal of cholestasis is 2 consecutive measurements of direct bilirubin < or = to 2mg/dL obtained at least 2 weeks apart.

SECONDARY OUTCOMES:
Essential fatty acid profile | Up to 30 days from therapy completion
  Previous studies have found no association between Omegaven administration and essential fatty acid deficiency. Due to theoretical concern for developing fatty acid deficiency with low dose Omegaven administration, these levels will be followed during Omegaven therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Sivan Kinberg, MD, MS, Principal Investigator — Columbia University
Locations (1):
- Columbia Presbyterian Medical Center-Children's Hospital of NY, New York, New York, United States